CLINICAL TRIAL: NCT02395146
Title: Intra-operative Monitoring of the External Branch of the Superior Laryngeal Nerve (EBSLN) During Thyroid Surgery: Does it Improve Voice Preservation?
Brief Title: Neural Monitoring of the Superior Laryngeal Nerve in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-04-06-SUR
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Laryngeal Nerve; Thyroid Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring (Experimental): intraoperative EBSLN monitoring will take place
  Interventions: Procedure: Monitoring
- Non-Monitoring (No Intervention): No intraoperative EBSLN monitoring will take place (standard practice)

INTERVENTIONS:
Procedure: Monitoring — intraoperative EBSLN monitoring
  Arms: Monitoring

SUMMARY:
Thyroid surgeons place an enormous amount of importance and rightly so to the preservation of the recurrent laryngeal nerve (RLN) during thyroidectomies. A good knowledge of the anatomy of the nerve and meticulous dissection technique and intraoperative identification of the nerve are crucial to the anatomic and functional integrity of the nerve. The use of intraoperative neural monitoring to aid the surgeon in the identification of the RLN has gained acceptance and is considered standard practice in several units. However, lesser emphasis has been placed historically on the identification and preservation of the external branch of the superior laryngeal nerve (EBSLN) during thyroid surgery. The EBSLN supplies the cricothyroid muscle that controls pitch variation during phonation. Unlike damage to the recurrent laryngeal nerve which manifests readily as vocal cord paralysis, intraoperative damage to EBSLN is difficult to assess postoperatively as visual assessment of the larynx is not indicative of the integrity of the nerve. Injury of the EBSLN can cause weakness or complete paralysis of the ipsilateral cricothyroid muscle. Patients may report a deeper voice or an inability to produce high pitched sounds.

Patients may also complain of weakness, tightness of the voice, and require extra effort to speak. Of note, voice changes with EBSLN injury are subtle in the general population but can be devastating in patients who depend on their voice for a living. Importantly, EBSLN injury is reported in upto 50% of thyroid surgery in contrast to 12% of recurrent laryngeal nerve injury during thyroid surgery. The new guidelines published in the Laryngoscope recommend routine intraoperative neural monitoring of EBSLN. The Investigators have a functional system in use currently for monitoring recurrent laryngeal nerve intraoperatively and propose to study the impact of monitoring the EBSLN using the same neural monitoring device to improve voice results following thyroid surgery.

DETAILED DESCRIPTION:
Thyroid surgery can result in change in the voice. This is because two nerves controlling the voice quality are situated very close anatomically to the thyroid gland and are at risk of damage during the surgery. One of the nerves that is called the recurrent laryngeal nerve controls the movements of the voice cords and is more readily identifiable and its injury is also detected easily by direct examination of the voice box as reduced/absent movement of the voice cord. It gets damaged in upto 1% of thyroid surgeries. The other nerve that is of interest to our study is called the superior laryngeal nerve, and its external branch (EBSLN) controls the pitch of the voice cord by supplying a muscle called the cricothyroid. This nerve is difficult to see and is reported to be damaged in 50% of thyroid surgeries. Its damage cannot be picked up on direct examination of the larynx and voice changes are subtle though devastating for individuals who depend on their voice for their livelihood singers actors etc. The Investigators would like to study if using a nerve monitor that is used to check the RLN during thyroid surgery can also be used to check the EBSLN. The Investigators hope that this could reduce the chances of damaging the nerve significantly. If the study shows good preservation of the EBSLN with the nerve monitor the Investigators will be able to make it a standard procedure during thyroid surgery.

The Investigators plan to recruit patients undergoing thyroid surgery involving one half of the thyroid gland. They will be given all the information about the study and consent will be obtained. If they agree to participate they will be divided into two groups randomly those who will have the intraoperative EBSLN monitoring and those who will not. All patients will have a preoperative voice assessment in the speech therapy unit which will involve filling in a voice questionnaire and undergoing a glottography (pitch assessment) They will then undergo the surgery Approximately 3 months after the surgery they will have another voice assessment using the voice questionnaire and the glottography. At this time they will also have an EMG assessment of the cricothyroid muscle which is the best method to check the function of the EBSLN. No further procedures/assessments will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic hemithyroidectomies (thyroid nodules 5 cm or less).
* age 18 and over
* able to provide informed consent

Exclusion Criteria:

* Patients who develop a recurrent laryngeal nerve palsy following surgery will be excluded from the study.
* Patients who withdraw consent during or after study
* Patients with pre-existing laryngeal pathology like reinkes edema, vocal cord nodules, laryngeal inflammation, previous laryngeal surgery etc
* Pregnant women (confirmed by history and routine pregnancy test)
* Those unable to give informed consent
* Previous major neck surgery such as neck dissections, laryngeal surgery, carotid endarterectomies, parathyroid and thyroid surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Intact external branch of the superior laryngeal nerve | 6 months
  Review and feedback via questionnaire of superior laryngeal nerve

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom